CLINICAL TRIAL: NCT06328153
Title: Biomechanically Based Fu's Subcutaneous Needling Treatment for Senile Keen Osteoarthritis: Protocol For a Randomized Controlled Trial
Brief Title: Efficacy and Mechanism of FSN Treatment for Senile Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jian Sun, Vice Dean of College, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BF2022-101
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Osteoarthritis; Fu's Subcutaneous Needling; Gait analysis; muscle elasticity
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSN group (Experimental): Fu's subcutaneous needling (FSN) is a new type of acupuncture. Patients in the FSN Group only received FSN treatment, without other interventions such as oral drugs or topical drugs.
  Interventions: Device: Fu's Subcutaneous Needling
- Drug Group (Active Comparator): Celecoxib is a member of Nonsteroidal Antiinflammatory Drugs (NSAIDs) and the most commonly used treatment for knee osteoarthritis. Patients in the drug group received only oral celecoxib, no other oral or topical drugs, and no other physical therapies.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Device: Fu's Subcutaneous Needling — Operation of the FSN will follow the KOA's Fu's Subcutaneous Needling Treatment Code of Practice24. After routine disinfection, a disposable Fu's subcutaneous needle ( Nanjing-Paifu Medical Technology Co., Ltd., Jiangsu, China ) is inserted parallel into the subcutaneous loose connective tissue of the pathological tight muscles ( gastrocnemius muscle, tibial anterior muscle and quadriceps femoris muscle ). The FSN needle is operated in a swaying movement. The fan angle is approximately 60°; perform a total of 45 round trips in 30 seconds. Swaying is accompanied by reperfusion approach: 20 sweeps with 10 seconds of reperfusion approach as a group, 3 groups for each pathological tight muscle. The reperfusion approach requires active, short and sharp contractions of the pathological tight muscle. The muscle alternates contraction and relaxation. The FSN group is treated 3 times a week for 2 weeks.
  Other Names: FSN; Fu's Subcutaneous Needling Treatment; FSN Treatment; Floating Needle; Floating Needle Treatment
  Arms: FSN group
Drug: Celecoxib — Participants in the drug group will receive celecoxib (capsule) 200mg every day continuously for 2 weeks.
  Other Names: Nonsteroidal Antiinflammatory Drugs; NSAIDs
  Arms: Drug Group

SUMMARY:
The goal of this clinical trial is to compare FSN with oral Nonsteroidal Antiinflammatory Drugs (NSAIDs) in pain relief and improvement in knee function among elder people, the main questions it aims to answer are:

Q1: Compared with the positive drug (celecoxib), whether FSN is more or at least as effective for pain relief and improvement in knee function in elder people with knee arthritis.

Q2: From the biomechanical point of view, what is the mechanism by which FSN plays a therapeutic role in knee osteoarthritis (KOA)?

Participants will:

1. Will be randomly assigned to 2 groups. There will be 30 participants in each group.
2. A group of patients will receive FSN monotherapy, while the other group will receive oral celecoxib and pantoprazole. Each patient will receive a 2-week course of treatment.
3. Visual analogue scale (VAS), WOMAC, knee range of motion (ROM), gait analysis, and musculoskeletal ultrasonography (US) of lower extremity muscles will be assessed during treatment and in the follow-up.

Researchers will compare FSN and celecoxib to see if FSN has better, or at least equivalent, efficacy than celecoxib, which is commonly used in clinical practice.

DETAILED DESCRIPTION:
This study was a randomised, parallel-controlled, single-center prospective clinical study, which included 60 participants, with an FSN group (n=30) and a drug group (n=30). All patients will give informed consent before participation and the trial is initiated after approval. The Fu's subcutaneous needling(FSN) group underwent FSN treatment 3 times a week for 2 weeks, while the drug group received oral celecoxib 0.2 g/day for 2 weeks, with a follow-up period of 2 weeks after the completion of treatment. The primary outcome will be the visual analog scale（VAS）after two weeks of treatment. The secondary outcomes will be self-reported knee stiffness using the WOMAC Index, joint active range of motion test, three-dimensional gait analysis, and Shear wave elastic imaging technology analysis in lower limb muscles. The results of this trial will be disseminated through publication in peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60-80 years old.
* BMI<28.
* Clinical diagnosis of knee osteoarthritis.
* Kellgren-Lawrence grade 1-3.
* Knee pain score > 3 on an 10-point numerical rating scale (VAS).
* Having no obvious deformity.
* Having not taken other medication and other modalities of treatment in the last 3 months.
* Voluntary and capable of signing the informed consent form.

Exclusion Criteria:

* Non-primary knee osteoarthritis, such as gouty arthritis and hemophilic arthritis, is caused by serious violence and the structure of the knee joint is damaged.
* Patients with other diseases that may cause lower limb pain, such as lumbar disc herniation and lumbar spinal stenosis.
* Patients with lower extremity vascular disease.
* Having a history of knee surgery in the past 6 months.
* Receiving drugs related to knee osteoarthritis or the internal and external treatment of traditional Chinese Medicine in the past 3 months.
* Severe systemic or lower limb local skin disease.
* Contraindications to NSAIDs, such as after coronary artery bypass grafting, active peptic ulcer, severe heart failure, etc.
* With any unstable medical or psychiatric illness.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the visual analogue scale (VAS) (0-100 mm) at the 14th day after receiving treatment. | Baseline and the 14th day after the start of treatment
  Visual analogue scale (VAS) is used to assess pain. A "0" indicates no pain or no limitation of function and gets worse as the value increases, and a "10" indicates severe pain (refractory to analgesic medication) or extreme limitation of function

SECONDARY OUTCOMES:
Change from Baseline in the visual analogue scale (VAS) (0-100 mm) at the 7th day, the 28th day and 42th day after the start of treatment. | Baseline and the 7th day, the 28th day and the 42th day after the start of treatment
  Visual analogue scale (VAS) is used to assess pain. A "0" indicates no pain or no limitation of function and gets worse as the value increases, and a "10" indicates severe pain (refractory to analgesic medication) or extreme limitation of function
Change from Baseline in The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index at the 7th day, the 14th day, the 28th day and 42th day after the start of treatment. | Baseline and the 7th day, the 14th day, the 28th day and the 42th day after the start of treatment.
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index is a scoring system that is applicable to the assessment of knee osteoarthritis. The severity of arthritis and the efficacy of treatment is evaluated according to the relevant symptoms and signs of patients. The rating scale includes 24 questions in 3 aspects of pain, stiffness and dysfunction, and there are 2 methods of calculation: 5-point scale (0-4) and 11-point scale (0-10), corresponding to a maximum score of 96 and 240, respectively. The higher the score, the more severe the subjective feeling of the symptoms.
Change from Baseline in the active range of motion (ROM) of the knee at the 7th day,the 14th day,the 28th day and 42th day after the start of treatment. | Baseline and the 7th day, the 14th day, the 28th day and the 42th day after the start of treatment
  A goniometer is used. In general, for healthy people, the active range of motion (ROM) of the knee joint is: extension-flexion (0°-135°). Limited flexion or extension of the knee, or a range beyond the normal range, may be the manifestation of knee disease.

OTHER OUTCOMES:
Change from Baseline in the data of the Three-dimensional gait analysis at the 7th day and 14th day after the start of treatment. | Baseline and the 7th day, the 14th day after the start of treatment
  The Opti_Knee 3D motion analysis system is used. Participants are made to walk continuously on the exercise board in a natural habitual position at a constant speed of 3.0km/h. The system collects gait data under appropriate working conditions, including six degrees of freedom data: femoral relative to tibial internal/external rotation angles, internal/external rotation angles, flexion/extension angles, anterior/posterior displacements, superior/inferior displacements, and internal/external displacements).The collected data help to analyze the mobility of the knee and even the whole lower limb.
Change from Baseline in the data of the shear wave elastic imaging technology analysis at the 7th day and 14th day after the start of treatment. | Baseline and the 7th day, the 14th day after the start of treatment
  Supersonic Colour Doppler Ultrasound Diagnostic Unit is used to detect and calculate the mean value of Young's modulus for the muscle tissues of the lower limb. Each frozen image is repeated 3 times, and the mean values of 2 qualified sampling boxes is taken for statistical analysis.
Incidence of Treatment-Emergent Adverse Events | Up to 6 weeks.
  Unfavourable or unintended events in participants in the study are documented using a pre-set questionnaire and appropriate management measures will be taken. If the subject develops a more serious adverse reaction and the investigator considers the subject unfit to proceed with the study, the trial will be terminated.

IPD SHARING:
Plan to Share IPD: Undecided
Details of individual participant data (IPD) sharing still need to be determined with institutional ethics committees.

REFERENCES:
- [Derived] Huang H, Liu R, Shao J, Chen S, Sun J, Zhu J. Biomechanically based Fu's subcutaneous needling treatment for senile knee osteoarthritis: protocol for a randomized controlled trial. J Orthop Surg Res. 2024 Jul 8;19(1):394. doi: 10.1186/s13018-024-04878-7. PMID 38978119